CLINICAL TRIAL: NCT00791063
Title: An Open-Label Study to Evaluate 18F ML-10 as a PET Imaging Radiotracer for Early Detection of Response of Brain Metastases to Whole Brain Radiation Therapy (WBRT)
Brief Title: 18F ML-10 for Early Detection of Response of Brain Metastases to WBRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aposense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NST-CA001CTIL
Record Dates: First submitted 2008-07-01; First posted 2008-11-14 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Solid Tumors; Brain Metastases
Keywords: cell death; Apoptosis; PET imaging; brain metastases; whole brain radiation therapy
MeSH Terms: conditions — Brain Neoplasms | interventions — 5-fluoropentyl-2-methylmalonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F ML-10 (Experimental): Intervention - 18F ML-10 PET/CT imaging for early detection of response of brain metastases to WBRT
  Interventions: Other: 18F ML-10

INTERVENTIONS:
Other: 18F ML-10 — Patients will undergo 2-3 brain PET/CT sessions; A pre-treatment session and 1-2 sessions post WBRT treatment. Each PET/CT session will be done following intravenous administration of 18F-ML-10, to assess tracer uptake by the tumor.
  Other Names: 18F ML-10 PET/CT imaging

SUMMARY:
The purpose of this study is to evaluate the potential of [18F]-ML-10 to serve as a non-invasive imaging tool for the early detection of apoptosis in brain metastases in response to radiation therapy. Such early detection may improve clinical management of patients with brain metastases, as it may help early identification of non-responders, and subsequently potentially lead to optimization of radiation dose, early decision on focal irradiation of selected, non-responsive lesions, or early referral of the patient to surgery. The experimental design of the present study aims to evaluate the potential of non-invasive PET examination with [18F]-ML-10, to provide the clinician early in the course of treatment, via non-invasive molecular imaging of radiation-induced apoptosis, information on tumor responsiveness, that is currently available only several weeks to months after completion of the radiotherapy.

DETAILED DESCRIPTION:
Early assessment of the efficacy of anti-cancer therapy is highly desirable and an unmet need in clinical oncology. Currently, treatment efficacy is mostly measured by following tumor size by anatomical imaging (CT scan or MRI). However, changes in tumor size may be observed only after several weeks to several months after completion of treatment. Meanwhile, in cases where there is no response, the patient is unnecessarily exposed to treatment's side effects, and precious time may be lost before the initiation of an alternative, potentially more beneficial line of therapy. Therefore, there is an urgent and serious need for better tools for monitoring of tumor response to anti-cancer treatments.

To address this need, [18F]-ML-10, a novel small molecular-weight probe (MW 205) was developed for clinical detection of apoptosis in vivo by positron emission tomography (PET). [18F]-ML-10 is a member of the ApoSense family of compounds, a novel class of molecular probes for molecular imaging of cell death. The first clinical indication for which [18F]-ML-10 is being developed is imaging of apoptosis in clinical oncology to monitor tumor response to radiation therapy.

Previous preclinical and clinical studies have substantiated the safety of [18F]-ML-10, its very high stability in vivo, its favorable biodistribution profile, and its efficacy in clinical detection of cell death. In preclinical studies, the selective retention of [18F]-ML-10 in the focus of the neurovascular cell death in cerebral ischemia was demonstrated in respective animal models. 18F-ML-10 has been examined in two clinical trials in Uppsala Imanet, Sweden, and has been found safe in administration to healthy subjects and to elderly subjects with acute ischemic cerebral stroke. In these clinical trials, [18F]-ML-10 was also found efficacious in the clinical imaging of apoptosis, being either physiological apoptosis as observed in the testes in young healthy males, and pathological cell death, as observed in the brains of patients with acute ischemic cerebral stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cancer, diagnosed as having brain metastases, wherein at least one of the tumors has the diameter of ≥ 1.5cm, as assessed by MRI or CT performed within 14 days prior to screening/enrollment.
2. Patients scheduled for WBRT.
3. Fully conscious patients who have been given written and verbal information, and have then provided informed consent.

Exclusion Criteria:

1. Unstable medical condition, such as ischemic heart disease, liver disease or pulmonary disease, which may risk the patient during the study, as judged by the investigator.
2. Renal failure, with serum creatinine > 1.5mg/dl.
3. Any known psychiatric disorder other than mild depression or anxiety.
4. Patients treated for diabetes mellitus either by oral hypoglycemic medications or insulin.
5. Allergy to any known medication or to any imaging agent, or allergy-originated diseases, as judged by the investigator.
6. Other condition that might jeopardize the safety of the patient or the evaluation of the study results, as judged by the investigator.
7. Treatment with any non-marketed investigational drug within 30 days prior to administration of [18F]-ML-10.
8. Current alcohol or drug abuse
9. Pregnancy or lactation.
10. Women of child-bearing potential who are not using an adequate and medically acceptable contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Assessment of a change in the uptake of [18F]- ML-10 by the tumor as observed in comparing the PET scans before and after WBRT. | 3 months

SECONDARY OUTCOMES:
Assessment of a relationship between the change in uptake of [18F]- ML-10 by the tumor, observed in the PET scans obtained during the study, and tumor shrinkage in response to treatment, as assessed by MRI or CT according to the RECIST criteria. | 3 months
Detection of a potential change in the uptake of [18F]- ML-10 by the healthy brain tissue, as observed in comparing the PET/CT scans before and after WBRT, reflecting potential damage to intact brain tissue, as an adverse effect of the irradiation. | 3 months
Assessment of the correlation between the PET/CT region of interest (ROI), delineated by [18F]-ML-10 imaging, and the corresponding anatomical imaging. | 3 months
Assessment of the safety of [18F]-ML-10 when administered to cancer patients undergoing WBRT. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Allen, M.D., Principal Investigator — Rabin Medical Center, Petach Tikva 49100, Israel